CLINICAL TRIAL: NCT04650867
Title: Non Invasive Characterization of Pediatric Inflammatory Bowel Diseases Using Multispectral Optoacoustic Tomography
Acronym: PED_MSOT_IBD
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 351_20B
Record Dates: First submitted 2020-11-17; First posted 2020-12-03 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2021-02

CONDITIONS: Crohn's Disease; Ulcerative Colitis; IBD
Keywords: MSOT; Crohn's Disease; Crohn Disease; CD; Ulcerative Colitis; UC; chronic inflammatory bowel disease; IBD
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Routine biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with Crohn's disease: Patients diagnosed or with suspected Crohn's disease.
  Interventions: Device: Multispectral Optoacoustic Tomography (MSOT)
- Patients with Ulcerative colitis: Patients diagnosed or with suspected Ulcerative colitis
  Interventions: Device: Multispectral Optoacoustic Tomography (MSOT)
- Patients with unclassified inflammatory bowel disease (U-IBD): Patients diagnosed or with suspected unclassified inflammatory bowel disease (U-IBD)
  Interventions: Device: Multispectral Optoacoustic Tomography (MSOT)

INTERVENTIONS:
Device: Multispectral Optoacoustic Tomography (MSOT) — Non-invasive transcutaneous MSOT imaging of the bowel wall (terminal ileum, ascending caecum/colon, transverse colon, descending colon, and sigmoid colon).

SUMMARY:
Monocentric, prospective observational study to assess bowel inflammation in children with chronic inflammatory bowel disease (IBD) using multispectral optoacoustic tomography (MSOT).

DETAILED DESCRIPTION:
Inflammatory bowel diseases (IBD) play a major role in child and adolescent medicine. 25 % of patients with IBD are younger than 18 years of age at diagnosis and 25 % of those are even younger than 10 years of age at disease onset. The incidence of IBD in children and adolescents is 5-11/100 000 in Germany. IBD comprises mainly two entities, namely Crohn's disease (CD) and ulcerative colitis (UC). Patients with CD develop chronic and intermittent transmural inflammation of the gastrointestinal tract, which manifests with symptoms like diarrhea, hematochezia, abdominal pain, fatigue and malnutrition. This often results in weight loss and an increased risk of numerous complications such as the development of fistulas, perforations and intestinal strictures. In addition, growth disturbances and delayed onset of puberty are more frequent. Overall, the course of the disease can only be compared between children and adults to a very limited extent, as the disease often progresses more rapidly and severely in children. Accordingly, the procedure and recommendations for children with CD differ from those of adults. In addition to clinical scores, laboratory chemical parameters (blood count, CrP, calprotectin) and imaging diagnostics (endoscopy, ultrasound, MRT) are available to assess disease activity. However, the latter are only of limited use for routine monitoring due to their invasiveness, the need for sedation and the use of contrast agents. Multispectral Optoacoustic Tomograph (MSOT) on the other hand allows, comparable to sonography, a non-invasive, quantitative imaging of the composition of target tissues in children without sedation. Previous studies have shown that the quantitative determination of hemoglobin provides information on blood flow and inflammatory activity in the bowel of adult patients with Crohn's disease. In this pilot study, the intestinal wall of children will be characterized by MSOT to differentiate between CD, UC, and unclassified inflammatory bowel disease (U-IBD) and to quantify changes and correlate them with routine parameters. This could lead to a new possibility of non-invasive evaluation of disease forms and activity comparable to previous findings in adult patients with CD.

ELIGIBILITY:
Inclusion Criteria:

1. CD patients

   * Diagnosis CD or suspected CD at initial diagnosis
   * Indication for endoscopy and sampling (biopsy)
2. UC patients

   * Diagnosis UC or suspected UC at initial diagnosis
   * Indication for endoscopy and sampling (biopsy)
3. U-IBD patients

   * Diagnosis U-IBD or suspected IBD at initial diagnosis
   * Indication for endoscopy and sampling (biopsy)

Exclusion Criteria:

* Pregnancy
* Nursing mothers
* Unstable patients: Need for continuous cardiopulmonary monitoring (ECG and pulse oximetry)
* Tattoo in the field of investigation
* Subcutaneous fat tissue over 3 cm
* Lack of written consent

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients from the Department of Pediatric and Adolescent Medicine, University Hospital Erlangen
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Quantitative amount of oxygenated/deoxygenated hemoglobin in a.u. | Single time point (1 day)
  Oxygenated/deoxygenated hemoglobin signals in the intestinal/bowel wall of children with different entities of IBD (CD vs. UC vs. U-IBD) derived by MSOT in arbitrary units (a.u.)

SECONDARY OUTCOMES:
Quantitative amount of fibrosis/collagen signal in a.u. | Single time point (1 day)
  fibrosis/collagen signals in the intestinal wall of children with different entities of IBD (CD vs. UC vs. U-IBD) derived by MSOT in arbitrary units (a.u.)
Quantitative amount of single wavelength signal in a.u. | Single time point (1 day)
  single wavelength signals in the intestinal wall of children with different entities of IBD (CD vs. UC vs. U-IBD) derived by MSOT in arbitrary units (a.u.)
Optoacoustic spectrum in a.u. | Single time point (1 day)
  Optoacoustic spectrum in the intestinal wall of children with different entities of IBD (CD vs. UC vs. U-IBD) derived by MSOT in arbitrary units (a.u.)
Endoscopic extent of inflammation | Single time point (1 day), +/- 7 days from MSOT Imaging
  Assessment of inflammation in endoscopies within different entities of IBD (CD vs. UC vs. U-IBD)
Histological extent of inflammation and fibrosis | Single time point (1 day), +/- 7 days from MSOT Imaging
  Assessment of inflammation and fibrosis in histological samples from biopsies within different entities of IBD (CD vs. UC vs. U-IBD)
Clinical evaluation | Single time point (1 day)
  Assessement of clinical disease status by PCDAI or PUCAI according to the CED within different entities of IBD (CD vs. UC vs. U-IBD)
Ultrasound | Single time point (1 day), +/- 1 day from MSOT Imaging
  Assessment of disease status by ultrasound within different entities of IBD (CD vs. UC vs. U-IBD)
Laboratory parameters (blood - c-reaktive protein (CrP)) | Single time point (1 day), +/- 7 day from MSOT Imaging
  Assessment of disease status by laboratory parameters (CrP) within different entities of IBD (CD vs. UC vs. U-IBD)
Laboratory parameters (stool - Calprotectin) | Single time point (1 day), +/- 14 day from MSOT Imaging
  Assessment of disease status by laboratory parameters (Calprotectin) within different entities of IBD (CD vs. UC vs. U-IBD)
MRI | Single time point (1 day), +/- 14 day from MSOT Imaging
  Assessment of disease status by MRI (if applicable) within different entities of IBD (CD vs. UC vs. U-IBD)

CONTACTS AND LOCATIONS:
Overall Officials: Ferdinand Knieling, MD, Principal Investigator — Department of Pediatric- and Adolescent Medicine, FAU Erlangen-Nürneberg
Locations (1):
- University Hospital Erlangen, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benchimol EI, Fortinsky KJ, Gozdyra P, Van den Heuvel M, Van Limbergen J, Griffiths AM. Epidemiology of pediatric inflammatory bowel disease: a systematic review of international trends. Inflamm Bowel Dis. 2011 Jan;17(1):423-39. doi: 10.1002/ibd.21349. PMID 20564651
- [Background] Rosen MJ, Dhawan A, Saeed SA. Inflammatory Bowel Disease in Children and Adolescents. JAMA Pediatr. 2015 Nov;169(11):1053-60. doi: 10.1001/jamapediatrics.2015.1982. PMID 26414706
- [Background] Sauer CG, Kugathasan S. Pediatric inflammatory bowel disease: highlighting pediatric differences in IBD. Med Clin North Am. 2010 Jan;94(1):35-52. doi: 10.1016/j.mcna.2009.10.002. PMID 19944797
- [Background] Assa A, Avni I, Ben-Bassat O, Niv Y, Shamir R. Practice Variations in the Management of Inflammatory Bowel Disease Between Pediatric and Adult Gastroenterologists. J Pediatr Gastroenterol Nutr. 2016 Mar;62(3):372-7. doi: 10.1097/MPG.0000000000000943. PMID 26284542
- [Background] Ruemmele FM, Veres G, Kolho KL, Griffiths A, Levine A, Escher JC, Amil Dias J, Barabino A, Braegger CP, Bronsky J, Buderus S, Martin-de-Carpi J, De Ridder L, Fagerberg UL, Hugot JP, Kierkus J, Kolacek S, Koletzko S, Lionetti P, Miele E, Navas Lopez VM, Paerregaard A, Russell RK, Serban DE, Shaoul R, Van Rheenen P, Veereman G, Weiss B, Wilson D, Dignass A, Eliakim A, Winter H, Turner D; European Crohn's and Colitis Organisation; European Society of Pediatric Gastroenterology, Hepatology and Nutrition. Consensus guidelines of ECCO/ESPGHAN on the medical management of pediatric Crohn's disease. J Crohns Colitis. 2014 Oct;8(10):1179-207. doi: 10.1016/j.crohns.2014.04.005. Epub 2014 Jun 6. PMID 24909831
- [Background] Turner D, Levine A, Escher JC, Griffiths AM, Russell RK, Dignass A, Dias JA, Bronsky J, Braegger CP, Cucchiara S, de Ridder L, Fagerberg UL, Hussey S, Hugot JP, Kolacek S, Kolho KL, Lionetti P, Paerregaard A, Potapov A, Rintala R, Serban DE, Staiano A, Sweeny B, Veerman G, Veres G, Wilson DC, Ruemmele FM; European Crohn's and Colitis Organization; European Society for Paediatric Gastroenterology, Hepatology, and Nutrition. Management of pediatric ulcerative colitis: joint ECCO and ESPGHAN evidence-based consensus guidelines. J Pediatr Gastroenterol Nutr. 2012 Sep;55(3):340-61. doi: 10.1097/MPG.0b013e3182662233. PMID 22773060
- [Background] Preiss JC, Bokemeyer B, Buhr HJ, Dignass A, Hauser W, Hartmann F, Herrlinger KR, Kaltz B, Kienle P, Kruis W, Kucharzik T, Langhorst J, Schreiber S, Siegmund B, Stallmach A, Stange EF, Stein J, Hoffmann JC; German Society of Gastroenterology. [Updated German clinical practice guideline on "Diagnosis and treatment of Crohn's disease" 2014]. Z Gastroenterol. 2014 Dec;52(12):1431-84. doi: 10.1055/s-0034-1385199. Epub 2014 Dec 4. No abstract available. German. PMID 25474283
- [Background] Dignass A, Preiss JC, Aust DE, Autschbach F, Ballauff A, Barretton G, Bokemeyer B, Fichtner-Feigl S, Hagel S, Herrlinger KR, Jantschek G, Kroesen A, Kruis W, Kucharzik T, Langhorst J, Reinshagen M, Rogler G, Schleiermacher D, Schmidt C, Schreiber S, Schulze H, Stange E, Zeitz M, Hoffmann JC, Stallmach A. [Updated German guideline on diagnosis and treatment of ulcerative colitis, 2011]. Z Gastroenterol. 2011 Sep;49(9):1276-341. doi: 10.1055/s-0031-1281666. Epub 2011 Aug 24. No abstract available. German. PMID 21866493
- [Background] Knieling F, Neufert C, Hartmann A, Claussen J, Urich A, Egger C, Vetter M, Fischer S, Pfeifer L, Hagel A, Kielisch C, Gortz RS, Wildner D, Engel M, Rother J, Uter W, Siebler J, Atreya R, Rascher W, Strobel D, Neurath MF, Waldner MJ. Multispectral Optoacoustic Tomography for Assessment of Crohn's Disease Activity. N Engl J Med. 2017 Mar 30;376(13):1292-1294. doi: 10.1056/NEJMc1612455. No abstract available. PMID 28355498
- [Background] Waldner MJ, Knieling F, Egger C, Morscher S, Claussen J, Vetter M, Kielisch C, Fischer S, Pfeifer L, Hagel A, Goertz RS, Wildner D, Atreya R, Strobel D, Neurath MF. Multispectral Optoacoustic Tomography in Crohn's Disease: Noninvasive Imaging of Disease Activity. Gastroenterology. 2016 Aug;151(2):238-40. doi: 10.1053/j.gastro.2016.05.047. Epub 2016 Jun 3. No abstract available. PMID 27269244